CLINICAL TRIAL: NCT04087265
Title: Accuracy of Trans Abdominal Ultrasound in Evaluating Bowel Preparation Adequacy Before Performing Colonoscopy
Brief Title: Accuracy of Trans-abdominal Ultrasound in Evaluating Bowel Preparation Adequacy Before Colonoscopy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The PI requested to terminate due to his schedule
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00222200
Record Dates: First submitted 2019-09-05; First posted 2019-09-12 (Actual); Last update posted 2020-11-04 (Actual); Status verified 2020-07

CONDITIONS: Bowel Preparation
Keywords: transabdominal ultrasound; bowel preparation; colonoscopy

STUDY DESIGN:
Masking Description: The endoscopist who performs the colonoscopy will be blinded to the ultrasound results.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Study Population (All Participants) (Other): Patients who are referring for scheduled screening colonoscopy
  Interventions: Diagnostic Test: Transabdominal ultrasound

INTERVENTIONS:
Diagnostic Test: Transabdominal ultrasound — Transabdominal ultrasound will be performed 30 minutes before colonoscopy

SUMMARY:
Adequate preparation of the large bowel is required for a successful colonoscopy. It has been reported that poor preparation exists in 25% of examinations, which may lengthen overall procedure time, lower adenoma detection rate, and lead to earlier repeated colonoscopy. Evaluating the large intestine preparation by transabdominal ultrasonography can be a helpful way to predict the quality of the colonoscopy before initiating the process and therefore prevent performing the procedure in case of inadequate preparation. Estimating the colon preparation using an easy, fast and low cost way as transabdominal ultrasound before performing the colonoscopy would help the physician determine the next step. In case of poor preparation, colonoscopy can be postponed and the patient can be saved from repeated colonoscopy. The aim of this is to determine the accuracy of transabdominal ultrasonography in evaluating bowel preparation adequacy before performing colonoscopy.

DETAILED DESCRIPTION:
Colonoscopy is the most effective method of visualizing the colon mucosa. Adequate bowel preparation, which leads to clear visualization of mucosal surface of the colon, is important for a successful colonoscopy. Studies have shown that inadequate bowel preparation increases the adenoma detection failure, decreases the accuracy, prolongs the procedure time, decreases surveillance intervals, increases costs and results in procedure related complications. Poor preparation affects as many as 25% of colonoscopies and leads to an increase cost of colonoscopies. Endoscopists have long struggled to find the most appropriate follow-up strategy when the quality of bowel preparation is suboptimal. There is evidence of surveillance overuse in low-risk patients as well as underuse in high-risk patients.

Using a non-invasive, low cost approach for evaluating the bowel preparation before initiating the colonoscopy can save the patient from additional costs and procedures. Sonography has been used as a method of evaluating bowel condition in some colorectal diseases, mostly in Crohn's disease. Advantages of using ultrasound are that it is widely available, none-invasive, does not require preparation and lacks radiation exposure.

Transabdominal bowel ultrasound has the potential to be used as a screening tool for evaluating bowel preparation adequacy before performing the colonoscopy. To the best of the investigators' knowledge this is the first study evaluating bowel preparation by means of sonography before performing colonoscopy.

Consent will be obtained from volunteer patients who agree with participating in the study. Demographic data will be collected about an hour before the procedure. Patients will undergo transabdominal ultrasound by a trained physician 30 minutes before the scheduled colonoscopy. All the ultrasounds will be performed by one person. The sonologist will perform transabdominal ultrasound evaluation of bowel preparation using the following tools and criteria:

The scale of intestinal lumen of each section will be classified into one of four types: (i) empty (no intraluminal content is observed and the lumen is contracted or emptied; small amount of gas in colon lumen can be pressed away from the region of interest by using the transducer); (ii) filled (the lumen is filled with fluid and no obvious solid content); (iii) retention (flatulence and/or content retention in the intestine, with no improvement after pressing on the abdomen or changing the position of the patient); and (iv) mixed (two or three of the conditions described above is observed at a single site, namely filled + empty, retention + empty, retention + filled or retention + filled + empty).

Evaluation criteria will be divided into two main groups: cleaning grade and cleaning range. For cleaning grade, the cleanliness of each section of the intestinal lumen is assigned to a grade according to the evaluation of the lumen, as just described: I = emptying; II = filled or filled + empty; III = I or II with some retention; and IV = complete retention. Grades I and II (clear display of the colon wall) will be termed "qualified". The qualified rate of bowel preparation will be calculated with the number of qualified sections divided by the total number of colon sections in the group. For cleaning range, patients will be divided into three classes according to the number of qualified colon sections: A = all seven colon sections are fully qualified; B = four to six sections are qualified; C = three or fewer are qualified.

The scheduled colonoscopy will be performed according to the standard of care and the bowel preparation will be assessed using the BBPS score* as a routine in all colonoscopies.

*:The Boston bowel preparation scale (BBPS) was developed to limit interobserver variability in the rating of bowel-preparation quality, while preserving the ability to distinguish various degrees of bowel cleanliness. Subjective terms, such as "excellent," "good," "fair," "poor," and "unsatisfactory," are replaced by a 4-point scoring system applied to each of the 3 broad regions of the colon: the right side of the colon (including the cecum and ascending colon), the transverse section of the colon (including the hepatic and splenic flexures), and the left side of the colon (including the descending colon, sigmoid colon, and rectum). The points are assigned as follows:

* 0, unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared.
* 1, portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid.
* 2, minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segment is seen well.
* 3, entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid.

ELIGIBILITY:
Inclusion Criteria:

* healthy adults referring for screening colonoscopy

Exclusion Criteria:

* pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-15 (Estimated); Primary Completion 2021-02 (Estimated); Study Completion 2021-03 (Estimated)

PRIMARY OUTCOMES:
Accuracy of transabdominal ultrasound in evaluating bowel preparation adequacy before colonoscopy as assessed by the Boston Bowel Preparation Scale (BPPS) | 4 months
  The BBPS was developed to limit interobserver variability in the rating of bowel-preparation quality, while preserving the ability to distinguish various degrees of bowel cleanliness. The points are assigned as follows:
  * 0 - unprepared colon segment with mucosa not seen because of solid stool that cannot be cleared.
  * 1 - portion of mucosa of the colon segment seen, but other areas of the colon segment are not well seen because of staining, residual stool, and/or opaque liquid.
  * 2 - minor amount of residual staining, small fragments of stool, and/or opaque liquid, but mucosa of colon segment is seen well.
  * 3 - entire mucosa of colon segment seen well, with no residual staining, small fragments of stool, or opaque liquid.
  The correlation between ultrasound score and BBPS score will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Anthony N Kalloo, MD, Principal Investigator — Johns Hopkins University

IPD SHARING:
Plan to Share IPD: No